CLINICAL TRIAL: NCT02382861
Title: A Prospective, Randomized and Controlled Study Estimating the Neurally Adjusted Ventilatory Assist (NAVA) Versus the Pressure Support Ventilatory (PSV) in Difficult Weaning From Mechanical Ventilation
Brief Title: Conventional vs Neurally Adjusted Ventilatory Assist in Difficult Weaning From Mechanical Ventilation
Acronym: SENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2012/12
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Failure
Keywords: Neurally adjusted ventilatory assist; Weaning; Mechanical ventilation; Extubation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVA group (Experimental): Management of the difficult weaning from mechanical ventilation by the NAVA.
  Interventions: Device: Neurally adjusted ventilatory assist
- Control group (Active Comparator): Conventional management of the difficult weaning from mechanical ventilation, with the pressure ventilation.
  Interventions: Device: Noninvasive pressure support ventilation

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist — In the NAVA group, the level of NAVA is daily adjusted to obtain Eadimax corresponding to 60 % of Eadimax of the patient during the SBT to obtain a good clinical and biologic tolerance, with a respiratory frequency between 15 and 30/min and a tidal volume at 6ml/kg.
  Arms: NAVA group
Device: Noninvasive pressure support ventilation — In the control group, the PSV is decreased of 2cmH2O daily or several times a day to obtain a good clinical and biologic tolerance, with a respiratory frequency between 15 and 30/min and a tidal volume at 6ml/kg.
  Arms: Control group

SUMMARY:
The NAVA, by its more physiological aspect and a better adaptation of the patient to the ventilator with a decrease of asynchronies patients-ventilators, could decrease the duration of weaning and so decrease the duration of invasive mechanical ventilation and the morbi-mortality. The objective of this study is to compare the neurally adjusted ventilatory assist versus the usual management of weaning from mechanical ventilation, in term of duration of weaning, at the patients in period of difficult weaning from the invasive mechanical ventilation.

DETAILED DESCRIPTION:
- Background: The NAVA is a new mode of ventilation which works from the continuous recording of the electromyogram of the diaphragm. In theory, the NAVA delivred a proportional and synchronous assistance, to respiratory efforts allowing a more adequate ventilatory support. However, no study estimates the NAVA in the weaning from mechanical ventilation.

- Purpose: The NAVA, by its more physiological aspect and a better adaptation of the patient to the ventilator with a decrease of asynchronies patients-ventilators, could decrease the duration of weaning and so decrease the duration of invasive mechanical ventilation and the morbi-mortality. The objective of this study is to compare the neurally adjusted ventilatory assist versus the usual management of weaning from mechanical ventilation, in term of duration of weaning, at the patients in period of difficult weaning from the invasive mechanical ventilation.

- Detailed description: Approximately 20 to 25 % of the patients under mechanical ventilation who have the general criteria of weaning will not pass a first SBT (Spontaneous Breathing Trial). At this moment, the management of the weaning ventilatoire are made with PSV. The NAVA is proportional assistance and depends on the intensity of the electric diaphragmatic signal (Edi). The respiratory effort of the patient is directly detected from the Edi signal. In theory, the NAVA is a proportional and synchronous respiratory.

* After a first failure of a SBT, patients respecting the inclusion criteria and exlusion criteria described above are then included in the study and randomized in two groups (control group or NAVA group).
* In the control group, the PSV is decreased of 2cmH2O daily or several times a day to obtain a good clinical and biologic tolerance, with a respiratory frequency between 15 and 30/min and a tidal volume at 6ml/kg.
* In the NAVA group, the level of NAVA is daily adjusted to obtain Eadimax corresponding to 60 % of Eadimax of the patient during the SBT to obtain a good clinical and biologic tolerance, with a respiratory frequency between 15 and 30/min and a tidal volume at 6ml/kg.
* Twice a day, the criteria of SBT are looked for. When they are present, a SBT is realized. If it is a success, the patient will be extube. If it is a failure, the patient will be reventilated in PSV or NAVA according to their group. A non-invasive ventilation preventive or of "rescue" can be administered post-extubation according to criteria. The reintubated criteria are also defined.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Under mechanical ventilation > 48 hours
* A first failure of a SBT
* Plateau pressure 30cmH2O with tidal volume 8ml / kg
* SpO2 ≥ in 90 % with a FiO2 ≥ 50 %, or PaO2 / FiO2 > 150mmHg
* Positive expiratory pressure 8cmH2O
* No more of one mg/hour of noradrenaline or adrenalin
* Temperature >36 and <39°C.
* Stable neurological state (Glasgow scale > 4) without sedation (or very low sedation).
* Consent, dated and signed by the patient or his representative.

Exclusion Criteria:

* Contraindications to the NAVA (recent high digestive suture or oesophageal varices bleeding < 4 days).
* Pregnant woman.
* Age <18 years.
* Tracheotomy.
* Cardiac arrest with a reserved neurological prognostic.
* Therapeutic limitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Duration of weaning from the mechanical invasive ventilation. | 48 hours after the extubation
  This duration is defined by the period between the first failure of the spontaneous breathing trial (SBT) and 48 hours after the extubation.

SECONDARY OUTCOMES:
Duration between the inclusion and the success of the SBT | 28th day
Duration of invasive mechanical ventilation | 28th day
Rate of failure of SBT | 28th day
Rate of success of SBT | 28th day
Rate of ventilator-associated pneumonia | 28th day
Length of intensive care unit stay | 28th day
Duration of hospitalization | 28th day

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, Doctor, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux Hôpital Pellegrin, Bordeaux, Aquitaine, France